CLINICAL TRIAL: NCT06394362
Title: Comparison of Deep Hypnotic Time Duration in Geriatric Patients Undergoing General Anesthesia With Additional Bispectral Index Monitoring Compared to Standard Monitoring at Cipto Mangunkusumo Hospital in 2023
Brief Title: Comparison of DHT Duration in Geriatric Patients Using BIS Monitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Riyadh Firdaus, MD, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: IndonesiaU230424
Record Dates: First submitted 2024-04-24; First posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Deep Hypnotic Time; Emergence Time; Geriatric Population; General Anesthesia
Keywords: bispectral index; deep hypnotic time; emergence time; mini mental state exam; geriatric population
MeSH Terms: interventions — Consciousness Monitors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental monitoring group with BIS (Experimental): Subjects who meet the study criteria and has signed the inform consent will be randomized in a 1:1 ratio into 2 groups, namely Group A undergoing general anesthesia with additional BIS monitoring. When the patient arrives in the preparation room approximately 1 hour before surgery, MMSE evaluation is conducted to obtain preoperative MMSE data. Before anesthesia induction, monitoring and BIS sensor placement are performed
  Interventions: Other: Bispectral index monitor
- Control monitoring group without BIS (No Intervention): Subjects who meet the study criteria and has signed the inform consent will be randomized in a 1:1 ratio into 2 groups, Group B undergoing general anesthesia with standard monitoring according to ASA. When the patient arrives in the preparation room approximately 1 hour before surgery, MMSE evaluation is conducted to obtain preoperative MMSE data. The BIS monitor for patients in Group B is then covered (hidden BIS), so that the data cannot be viewed by the anesthesia team performing the anesthesia

INTERVENTIONS:
Other: Bispectral index monitor — Bispectral Index (BIS), that was introduced in 1992, is a tool that monitors the depth level of hypnosis through data processing of an electroencephalogram using computer algorithm and presented in the form of processed EEG. Utilizing BIS as a monitoring tool has shown effectiveness in reducing recovery time, prevent awareness, and bring down the amount of anesthesia agent however, as of now, it has not been incorporated into the 2020 American Society of Anesthesiologists (ASA) standard procedure on anesthesia monitoring. aims to comparing the deep hypnotic time duration on two group of geriatric patients which undergoes general anesthesia with BIS monitoring compared to standard monitoring.
  Arms: Experimental monitoring group with BIS

SUMMARY:
Without adequate monitoring, administration of anesthetic agents can create unnecessary deeper anesthetic plane in geriatric population. This study aims to compare the duration of deep hypnotic time (DHT) in geriatric patients undergoing general anesthesia with additional BIS monitor compared to standard monitoring. This study was a randomized clinical trial involving 44 geriatric patients undergoing general anesthesia. Subjects are divided into two groups, one with additional BISTM monitor and the other with standard monitoring. Data acquired from BISTM will continually be recorded to be analyzed afterward

ELIGIBILITY:
Inclusion Criteria:

* Sampling was consecutively conducted on geriatric patients aged >60 years undergoing general anesthesia for procedures lasting >2 hours with ASA physical status 1-3 and willing to participate in the study

Exclusion Criteria:

* Exclusion criteria included intracranial procedures, unstable hemodynamic conditions, neurocognitive impairment, and if the patient was anticipated not to be extubated at the end of the surgical procedure. Patients could be excluded if the preoperative MMSE score was <24, undergoing general anesthesia using a combination of ketamine and/or N20 agents, experiencing emergencies during surgery, and losing BIS data >10% of the duration of the operation

Ages: 61 Years to 71 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-02-10 (Actual)

PRIMARY OUTCOMES:
Deep Hypnotic time duration with Bispectral Index Monitoring | 24 hours
  Deep Hypnotic Time is the period during the Bispectral Index (BIS) are extensively less than 40 (a scale of 0 - 100). The BIS value that is believed to prevent 50% of the population from responding to verbal instructions placed on an index value of 67 - 79. Targeted BIS value to prevent awareness under general anesthesia are at a range of 40 - 60. A study conducted using BIS, shows that under a standard care, BIS value during operative maintenance period tends to be lower which sat around 36 (31 - 49). Duration is the lower the DHT duration the better the outcome of the patient, duration is measured in minutes

SECONDARY OUTCOMES:
Mini Mental State Examination exam before and after operation in both control and experimental group | 24 hours
  patients mental state is examined by using MMSE test to find an objective screening method of cognitive function (lost score = 0, maximum score = 40), scoring category : 0 - 10 MMSE Score = Severe Cognitive Impairment 10 - 20 MMSE Score = Moderate Cognitive Impairment 20 - 25 MMSE Score = Mild Cognitive Impairment 25 - 30 MMSE Score = Questionably Significant / Maybe Normal Cognitive

CONTACTS AND LOCATIONS:
Locations (1):
- Cipto Mangunkusumo Central National Hospital, Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided